CLINICAL TRIAL: NCT00041054
Title: A Phase II Study of Carboplatin, Etoposide, and Exisulind in Patients With Extensive Small Cell Lung Cancer
Brief Title: Combination Chemotherapy and Exisulind in Treating Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-30104; CLB-30104; CDR0000069439 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Etoposide; sulindac sulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carboplatin + etoposide + exisulind (Experimental): Patients receive carboplatin IV over 30 minutes on day 1 and etoposide IV over 30-60 minutes on days 1-3. Patients also receive oral exisulind twice daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months for 1 year and then every 4 months for 2 years.
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: exisulind

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Drug: exisulind

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Exisulind may make tumor cells more sensitive to chemotherapy. Combining chemotherapy with exisulind may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy with exisulind in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the percentage of patients with extensive stage small cell lung cancer who live more than 12 months after treatment with carboplatin, etoposide, and exisulind.
* Determine the response rate of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV over 30 minutes on day 1 and etoposide IV over 30-60 minutes on days 1-3. Patients also receive oral exisulind twice daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 4 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Lesions considered nonmeasurable include:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions situated in a previously irradiated area
* Must not be considered for combined chemotherapy and radiotherapy
* No active CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST no greater than 2 times ULN
* No clinically significant hepatic disease

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No clinically significant renal disease

Cardiovascular:

* No clinically significant cardiac disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent uncontrolled illness
* No known sensitivity to sulindac

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy for small cell lung cancer
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal agents except:

  * Steroids for adrenal failure
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent use of dexamethasone as an antiemetic

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy, including for palliation
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* More than 7 days since prior sulindac
* No concurrent sulindac

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-06; Primary Completion 2004-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
percentage of patients with extensive stage small cell lung cancer who live more than 12 months after treatment | Up to 3 years

SECONDARY OUTCOMES:
response rate | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, MD, Study Chair — Washington University Siteman Cancer Center
Locations (83):
- United States (81):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- McGill University, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Govindan R, Wang X, Baggstrom MQ, Burdette-Radoux S, Hodgson L, Vokes EE, Green MR; Cancer and Leukemia Group B. A phase II study of carboplatin, etoposide, and exisulind in patients with extensive small cell lung cancer: CALGB 30104. J Thorac Oncol. 2009 Feb;4(2):220-6. doi: 10.1097/JTO.0b013e3181951eb0. PMID 19179900
- [Derived] Hanna M, Thipphawong J; 118 Study Group. A randomized, double-blind comparison of OROS(R) hydromorphone and controlled-release morphine for the control of chronic cancer pain. BMC Palliat Care. 2008 Oct 31;7:17. doi: 10.1186/1472-684X-7-17. PMID 18976472